CLINICAL TRIAL: NCT01656681
Title: A 64-week Pilot Trial to Evaluate the Effects of a Novel Nutraceutical on Weight Loss and Weight Loss Maintenance in Obese Subjects
Brief Title: Effect of a Novel Nutraceutical on Weight Loss and Weight Maintenance in Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MetaProteomics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: WLM1-FMR-CT
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- THIAA (Experimental): Stage 1 (the first 12 weeks of the study): all subjects participate in a structured lifestyle change program featuring a high-protein, high-phytonutrient food plan (HP2). Those randomized to THIAA arm additionally receive the THIAA tablet, 3 times a day.
  Stage 2 (the subsequent 52-week study): All qualified subjects (i.e. those who have lost at least 7.5% of their body weight in Stage 1) participate in a less restrictive lifestyle change program featuring a Mediterranean-style Low-glycemic-load food plan (MLGL). Those randomized to THIAA arm additionally receive the THIAA tablet, 3 times a day.
  Interventions: Dietary Supplement: THIAA
- Placebo (Active Comparator): Stage 1 (the first 12 weeks of the study): all subjects participate in a structured lifestyle change program featuring a high-protein, high-phytonutrient food plan (HP2). Those randomized to Placebo arm receive the placebo tablet, 3 times a day.
  Stage 2 (the subsequent 52-week study): All qualified subjects (i.e. those who have lost at least 7.5% of their body weight in Stage 1) participate in a less restrictive lifestyle change program featuring a Mediterranean-style Low-glycemic-load food plan (MLGL). Those randomized to Placebo arm receive the placebo tablet, 3 times a day.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: THIAA — A tablet containing 400 mg tetrahydro iso-alpha acids, 3 times a day
  Arms: THIAA
Dietary Supplement: Placebo — Placebo tablet
  Arms: Placebo

SUMMARY:
The purpose of this 2-stage intervention study is to investigate the effect of a novel nutraceutical (containing tetrahydro iso-alpha acids derived from hops) on weight loss and weight loss maintenance in obese participants.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30 and ≤ 47

Exclusion Criteria:

* Prohibited medications, supplements or herbal products

  1. Use of narcotics, oral or injectable corticosteroids, multivitamin/multimineral supplements, antioxidant supplements, vitamin D supplements, probiotics and omega-3 fatty acid supplements 30 days prior to screening and for the duration of the study.
  2. Use of prescription medications and/or nonprescription medications for acute medical conditions, semi-acute medical conditions, and weight loss.
  3. Change in prescription, OTC, nutritional supplements and or medical foods within 30 days prior to the beginning of the study and for the duration of the study.
* Medical history and concurrent diseases

  1. Known allergy or hypersensitivity to study product or placebo.
  2. Clinically significant abnormalities in medical history of physical examination.
  3. Clinically relevant conditions expected to preclude achievement of exercise recommendation.
  4. Hepatic, renal, gastrointestinal, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, or hematologic disease.
  5. Diabetes mellitus, irritable bowel syndrome, Gastro-esophageal reflux disease, HIV, TB ,hepatitis B or C, malignancy, sleep apnea, insomnia (requiring use of sleeping medication more than once weekly), night eating syndrome, Anorexia nervosa, bulimia, of non-specific eating disorder, and serious psychiatric illness.
  6. Smoking or use of nicotine containing products within 30 days prior to screening and for the duration of the study.
  7. Use of drugs of abuse (e.g. marijuana, cocaine, PCP, and methamphetamine) within 30 days prior to screening and for the duration of the study.
* Other criteria

  1. Initiation of a new or change of an existing exercise regiment within 30 days prior to screening.
  2. Initiation of a new or change of an existing food plan within 30 days prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Weight loss maintenance | Baseline, 64 weeks
  The primary endpoint is the absolute pounds of weight change from baseline to the end of the 64 weeks.

SECONDARY OUTCOMES:
Weight loss | Baseline, 12 weeks
  Percent weight loss at the end of 12 weeks (i.e. the Stage 1 of the trial where subjects participate in HP2).
Weight loss | Baseline, 12 weeks
  Absolute amount of weight loss at the end of 12 weeks (i.e. the Stage 1 of the trial where subjects participate in HP2).
Short-term THIAA effect | Baseline, 12 weeks
  Comparing the difference in absolute amount of weight loss between 2 arms at the end of 12 weeks (i.e. the Stage 1 of the trial).
Short-term THIAA effect | Baseline, 12 weeks
  Comparing the difference in percent weight loss between 2 arms at the end of 12 weeks (i.e. the Stage 1 of the trial).
Weight loss | 12 weeks, 64 weeks
  To evaluate absolute amount of weight loss during Stage 2 of the trial where subjects participate in MLGL (i.e. 12 weeks to 64 weeks).
Weight loss | 12 weeks, 64 weeks
  To evaluate percent weight loss during Stage 2 of the trial where subjects participate in MLGL (i.e. 12 weeks to 64 weeks).
Long-term THIAA effect | baseline, 64 weeks
  To evaluate the difference between 2 arms the amount of weight loss during the trial (i.e. baseline to 64 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Lamb, MD, Principal Investigator — MetaProteomics / Metagenics
Locations (1):
- Functional Medicine Research Center, Gig Harbor, Washington, United States